CLINICAL TRIAL: NCT07367386
Title: Evaluating the Impact of Increasing BMI on the Success of Neuraxial Blocks in Class III Obese Parturients: A Retrospective Cohort Study
Brief Title: Impact of Increasing BMI on the Success of Neuraxial Blocks in Class III Obese Parturients
Status: Completed | Type: Observational
Sponsor: Mariah Arif (Other Government)
Responsible Party: Sponsor-Investigator, Mariah Arif, Resident Physician, Hamad General Hospital
Organization: Hamad General Hospital (Other Government)
Other Study IDs: MRC-01-24-905
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Neuraxial Blocks
Keywords: Neuraxial blocks; Obesity; Parturient; Cesarean
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Class III obese parturient: Class III obese parturient undergoing cesarean section under neuraxial block
  Interventions: Procedure: Neuraxial anesthesia

INTERVENTIONS:
Procedure: Neuraxial anesthesia — Single-shot spinal anesthesia
Procedure: Neuraxial anesthesia — Epidural anesthesia
Procedure: Neuraxial anesthesia — Combined spinal-epidural anesthesia

SUMMARY:
This study seeks to compare the success rates, feto-maternal outcomes, and complications associated with different neuraxial blocks in Class III obese parturient undergoing cesarean section

DETAILED DESCRIPTION:
This was a retrospective cohort study. The data was obtained from electronic medical records of the eligible participants.

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal to 18 years
* BMI ≥ 45 kg/m²
* Gestational age ≥ 28 weeks

Exclusion Criteria:

* Age < 18 years
* BMI < 45 kg/m²
* History of venous thromboembolism or arterial disease (e.g., DVT, PE, angina, MI, or stroke)
* Severe active lung, cardiovascular, renal, or liver disorders; autoimmune disease; or hemoglobinopathies
* Hereditary or acquired thrombophilia (e.g., Factor V Leiden mutation or antithrombin deficiency)
* In utero fetal demise (IUFD)
* Failed operative vaginal delivery
* Cesarean for the second twin or multiple pregnancies (triplets or higher)
* IVF pregnancy
* Intraoperative bleeding>1500mL
* Emergency cesarean section (Category I)
* Presence of large uterine fibroid ≥10 cm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Study Population: Class III Obese parturients undergoing C-section under neuraxial blocks in the operating rooms of Women's Wellness and Research Center from 1 January 2025 to 1 December 2024.
Sampling Method: Non-Probability Sample
Enrollment: 1917 (Actual)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Failed neuraxial block | From onset of block until surgery completion
  Determine the occurrence of the conversion to general anesthesia

SECONDARY OUTCOMES:
Maternal adverse events | From onset of blockade until surgery completion
  Determine the incidence of maternal hypotension, bradycardia, high-spinal (above T1 level), level of blockade higher than T4, post-dural puncture headache
Fetal outcomes | At one and five minutes after birth
  Apgar score

CONTACTS AND LOCATIONS:
Overall Officials: Ayten Saracoglu, Principal Investigator — University of Florida, UF Health, Jacksonville, FL 32209, USA
Locations (1):
- Women's Wellness and Research Center, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No